CLINICAL TRIAL: NCT05751031
Title: Pregnancy and Neonatal Outcomes Following Antenatal Exposure to Raltegravir: a Pooled Analysis From the European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Penta UK (Network)
Collaborators: UCL Great Ormond Street Institute of Child Health (Other)
Responsible Party: Sponsor
Organization: PENTA Foundation (Network)
Other Study IDs: Raltegravir
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC): Pregnant women living with HIV and their infants from 9 European cohorts and studies within the European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir exposure in pregnant women living with HIV in routine clinical care. No study intervention administrated.

SUMMARY:
Raltegravir is the preferred INSTI for for treatment of antiretroviral-naïve pregnant women in the US Perinatal Guidelines, alongside Dolutegravir, and for late pregnancy. There are relatively limited information available on its use during early pregnancy, particularly the peri-conception period. The aim of the study is to assess "real-world" maternal, fetal and newborn outcomes following RAL use during pregnancy through pooled analysis of individual patient data from observational studies participating in the European Pregnancy and Paediatric Infections Cohort Collaboration.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women living with HIV, exposed to Raltegravir at any time during the pregnancy participating in EPPICC and their infants.

Exclusion Criteria:

* see inclusion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women with any exposure to RAL at any time during the pregnancy and their infants will be included in the analysis. With respect to eligibility, we will include any pregnancy reported within the participating studies with any RAL exposure regardless of pregnancy outcome, including those where the pregnancy is still ongoing at the time of the data merger. This analysis will be based on two EPPICC data mergers, one collecting data on eligible pregnancies with estimated date of delivery prior to 2015, and the second collecting data on eligible pregnancies since 2015 (2020/2021 merger).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Patterns of antenatal use | 12 months
  To describe patterns of antenatal use of RAL-containing regimens, including maternal characteristics, timing of initiation, NRTI backbone/other drugs in regimen and calendar time trends
Frequency of averse birth outcomes | 12 months
  To describe the frequency of adverse birth outcomes in RAL-exposed pregnancies including birth defects, stillbirths, preterm births, low birth weight infants, and small-for-gestational age infants, by timing of exposure
Birth defects per trimester of exposure | 12 months
  To compare risk of birth defects in infants with peri-conception and/or first trimester exposure to RAL with that in infants with exposure to RAL from the second or third trimester

SECONDARY OUTCOMES:
Frequency of discontinuation | 12 months
  To assess the frequency of discontinuation of RAL during pregnancy and potential reasons where data are available.
Viral suppression | 12 months
  To describe the proportion of women on RAL who achieve viral suppression by the end of pregnancy and the vertical transmission rate in mother-infants pairs with RAL use

CONTACTS AND LOCATIONS:
Overall Officials: Claire Thorne, Study Chair — Professor of infectious disease epidemiology
Locations (10):
- Centre Hospitalier Universitaire Saint Pierre, Brussels, Belgium
- Università degli studi di Firenze, Florence, Italy
- "Victor Babes" Hospital, Bucharest, Romania
- Russia (3):
  - State Budgetary Institution of Health Protection Irkutsk, Arkhangelsk
  - St Petersburg Republican Hospital, Saint Petersburg
  - St. Petersburg State Budgetary Health Institution, Saint Petersburg
- Spain (2):
  - Hospital San Joan de Deu, Barcelona
  - Hospital Clinico San Carlos, Madrid
- University Hospital Zurich, Zurich, Switzerland
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No